CLINICAL TRIAL: NCT07328698
Title: Effect of Postoperative Ozonated Oil Dressing on Early Wound Inflammation After Open Mesh Inguinal Hernia Repair: A Prospective Randomized Pilot Controlled Trial
Brief Title: Postoperative Ozonated Oil Dressing After Open Inguinal Hernia Repair: A Randomized Pilot Trial
Acronym: OZONE-HERNIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Alirıza Erdoğan, Medical doctor, General surgery, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/140
Record Dates: First submitted 2025-12-27; First posted 2026-01-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Inguinal Hernia Unilateral; Postoperative Wound Inflammation
Keywords: Inguinal hernia repair; Open inguinal hernia surgery; Ozonated oil; Ozonated oil dressing; Postoperative wound inflammation; Surgical wound care; Topical ozone; Pilot randomized controlled trial; Clean surgical wound; Wound surface temperature

STUDY DESIGN:
Intervention Model Description: This is a single-center, two-arm, parallel-group randomized pilot trial with 1:1 allocation to ozonated oil dressing versus standard sterile dressing after elective open mesh inguinal hernia repair, with follow-up through postoperative day 30.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Surgeons and clinical staff applying the dressing are not blinded due to the nature of the intervention and the characteristic odor of ozonated oil. Participants are not informed of group allocation and are unable to distinguish the dressing content. Outcome assessors, wound photograph evaluators, and statisticians are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozonated Oil Dressing (Experimental): Participants receive a sterile gauze dressing impregnated with CE-certified ozonated oil applied to the surgical incision after skin closure. The dressing is changed once daily for the first 48 hours, followed by standard wound care.
  Interventions: Drug: ozonated oil
- Standard Sterile Dressing (Active Comparator): Participants receive a standard sterile dry dressing applied to the surgical incision after skin closure. The dressing is removed within 24-48 hours postoperatively, and subsequent wound care is continued according to routine institutional practice.
  Interventions: Other: Standard Sterile Dressing

INTERVENTIONS:
Drug: ozonated oil — Ozonated oil-impregnated sterile gauze is applied topically to the surgical incision immediately after skin closure. The dressing is changed once daily for the first 48 hours postoperatively, followed by standard wound care according to institutional routine.
  Arms: Ozonated Oil Dressing
Other: Standard Sterile Dressing — A standard sterile dry dressing is applied to the surgical incision after skin closure and removed within 24-48 hours postoperatively. Subsequent wound care is continued according to routine institutional practice.
  Arms: Standard Sterile Dressing

SUMMARY:
This study looks at whether a special wound dressing containing ozonated oil can reduce early wound inflammation after open inguinal hernia surgery. Open inguinal hernia repair is a common operation, and although infection rates are low, many patients experience redness, swelling, tenderness, or discomfort at the surgical site during the first days after surgery.

Participants undergoing elective open inguinal hernia repair will be randomly assigned to receive either an ozonated oil-impregnated dressing or a standard sterile dressing after the operation. The main outcome is the level of wound inflammation measured on the third day after surgery. Other outcomes include wound temperature, pain levels, cosmetic healing, and wound-related problems during the first 30 days.

The ozonated oil used in this study is a CE-certified medical product that is already used in routine wound care. This pilot study aims to provide preliminary data to help determine whether ozonated oil dressing may improve early wound healing compared with standard care.

DETAILED DESCRIPTION:
Early postoperative wound inflammation following open inguinal hernia repair may affect patient comfort, recovery experience, and cosmetic outcome, even in the absence of surgical site infection. Although open mesh inguinal hernia repair is classified as clean surgery, localized inflammatory findings such as erythema, edema, tenderness, and increased wound temperature are commonly observed during the early postoperative period.

Ozonated oil is a CE-certified topical medical product that has been used in routine clinical practice for wound care in dermatology, plastic surgery, and chronic wound management. Its proposed mechanisms include antimicrobial activity, modulation of local inflammatory response, and support of tissue repair. However, randomized evidence evaluating its effect on early inflammatory response in clean elective surgical incisions remains limited, and most existing studies rely primarily on subjective assessments.

This single-center, prospective, randomized pilot controlled trial is designed to compare ozonated oil-impregnated dressing with standard sterile dressing after elective open inguinal hernia repair. The study focuses on early wound inflammation rather than infection as the primary endpoint, using a composite clinical and photographic inflammation score assessed by blinded evaluators. Objective assessment of local inflammation is supported by non-contact infrared wound surface temperature measurement.

Due to the low expected incidence of surgical site infection in this surgical setting, the study is not powered to detect statistically significant differences in infection rates. Infection-related outcomes are therefore collected for exploratory purposes only. As a pilot trial, the primary aim is to generate preliminary data on feasibility, effect size, and outcome variability to inform the design of future larger-scale randomized studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years
* ASA physical status I-III
* Scheduled for elective, unilateral open inguinal hernia repair
* Able to provide written informed consent

Exclusion Criteria:

* Emergency inguinal hernia (incarcerated or strangulated)
* Recurrent inguinal hernia
* Concomitant surgical procedures during the same operation
* Immunosuppression or long-term systemic steroid use
* Use of anticoagulant or antiplatelet therapy
* Known bleeding disorders
* Active dermatologic disease at the surgical incision site
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Composite Wound Inflammation Score | Postoperative day 3
  A composite wound inflammation score ranging from 0 to 12, consisting of erythema, edema, and exudate graded from standardized wound photographs (0-3 points each) and wound tenderness assessed during clinical examination (0-3 points). Wound photographs are independently evaluated by two blinded surgeons.

SECONDARY OUTCOMES:
Wound Surface Temperature Difference | Postoperative day 3
  Difference between mean surgical wound surface temperature and contralateral symmetrical skin temperature measured using a non-contact infrared thermometer.
Postoperative Pain Score | 6 hours, 24 hours, and postoperative day 3
  Pain intensity at the surgical site measured using a 0-10 visual analog scale (VAS).
Cosmetic Outcome Score | Postoperative day 30
  Patient-reported cosmetic satisfaction assessed using a 0-10 visual analog scale and photographic evaluation using the Hollander Wound Evaluation Score.
Surgical Site Infection | Within 30 postoperative days
  Incidence of surgical site infection defined according to Centers for Disease Control and Prevention (CDC) criteria, collected for exploratory analysis.
Additional Antibiotic Use or Unplanned Healthcare Visits | Within 30 postoperative days
  Any wound-related antibiotic treatment or unplanned medical visits due to wound complications during the postoperative follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rıza Erdoğan, Medical doctor, Principal Investigator — Private practice office
Locations (1):
- Dr. Ali Rıza Erdoğan Private Practice Office, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this is a single-center pilot study with a small sample size, and the dataset includes clinical and photographic wound data that could pose a risk of re-identification. Data sharing was not planned at the time of study design.